CLINICAL TRIAL: NCT00003591
Title: A Phase II Trial of External Irradiation (50.4 GY) and Weekly Paclitaxel (Taxol) for Non-Metastatic, Unresectable Pancreatic Cancer
Brief Title: Radiation Therapy Plus Paclitaxel in Treating Patients With Nonmetastatic, Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9812; CDR0000066661
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pacilitaxel + External Beam Radiation Therapy (PXRT) (Experimental): Paclitaxel 50 mg/m2 given on Days 1, 8, 15, 22, 29 and 36. Radiation therapy: 50.4 Gy/28 fractions (1.8 Gy per fraction) once a day in 5.5 weeks.
  Interventions: Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy plus paclitaxel in treating patients who have nonmetastatic, unresectable pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate of patients with nonmetastatic, unresectable pancreatic cancer receiving external beam irradiation and weekly paclitaxel. II. Determine the median survival after this treatment in these patients. III. Evaluate the acute and late treatment morbidity of paclitaxel in these patients. IV. Correlate p53 status with treatment response to this treatment in this patient population.

OUTLINE: This is a open label, multicenter study. Patients are highly recommended to undergo laparoscopic surgical staging prior to protocol to exclude peritoneal and hepatic metastases. Patients receive paclitaxel IV over 3 hours weekly for 6 weeks beginning on day 1 followed 1.5 hours later by external beam radiotherapy daily 5 days a week for 5.5 weeks beginning on day 1. All patients are restaged with an abdominal CT scan 6 weeks following completion of chemoradiotherapy. If there is marked response to treatment at this time, curative surgery may be attempted at the discretion of the attending surgeon. Patients are followed every 3 months for 1 year, every 4 months for the second year, every 6 months for years 3-5, and annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients will be accrued into this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed nonmetastatic, unresectable pancreatic adenocarcinoma No evidence of metastatic disease in the major viscera and no peritoneal seeding Residual disease after resection (R-1 or -2 micro- and macroscopic residual) eligible if measurable disease on the post operative CT or MRI scan Recurrent disease following radical surgery is eligible All malignant disease must be encompassable within a single irradiation field Must be a radiographically assessable disease CT with 5 mm cuts or spiral CT

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,800/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL Biliary system stented Renal: Creatinine less than 3.0 mg/dL OR Creatinine clearance at least 40 mL/min Other: If patients have biliary or gastroduodenal obstruction, they must have drainage prior to starting chemoradiation Oral intake of at least 1,500 calories per day No significant infection or other coexistent medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior paclitaxel At least 4 weeks since prior gemcitabine No other prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy to the planned field Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 1998-11; Primary Completion 2001-06 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To determine the one-year and median survival rates after PXRT
  To determine the one-year and median survival rates after paclitaxel and external beam radiation therapy (PXRT)

SECONDARY OUTCOMES:
To determine the response rate of PXRT in unresectable pancreatic cancer in a multi-center trial
To evaluate the acute and late treatment morbidity of paclitaxel in a multi-institutional setting
To correlate p53 status with treatment response to PXRT

CONTACTS AND LOCATIONS:
Overall Officials: Tyvin A. Rich, MD, Study Chair — University of Virginia
Locations (234):
- United States (218):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Urology Associates - Mobile AL, Mobile, Alabama
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Cancer Therapy Center, Anchorage, Alaska
  - Arizona Cancer Center, Tucson, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Mount Diablo Medical Center, Concord, California
  - Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Kaiser Permanente Medical Center - Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Cancer Care Center, Pomona, California
  - Mercy Medical Center - Redding, Redding, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Santa Cruz Radiation Oncology Medical Group, Inc., Santa Cruz, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Stanford University, Stanford, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Radiation Oncology Center - Walnut Creek, Walnut Creek, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Whittingham Cancer Center, Norwalk, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - West Florida Cancer Institute - Pensacola, Pensacola, Florida
  - Bayfront Medical Center, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - St. Joseph's Radiation Oncology Center, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Medical Center at Bowling Green, Bowling Green, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Western Baptist Hospital, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Joint Center for Radiation Therapy, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - Veterans Affairs Medical Center - Saint Louis, St Louis, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Elizabeth General Medical Center - West, Elizabeth, New Jersey
  - South Jersey Hospital - Millville, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua-Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Kaplan Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - Genesee Hospital - Rochester, Rochester, New York
  - University of Rochester Cancer Center, Rochester, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - UNI-MED Medical Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Samaritan Regional Cancer Center, Corvallis, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Penn State Geisinger Medical Center, Danville, Pennsylvania
  - Mercy Catholic Medical Center, Mercy Fitzgerald Divison, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Allegheny University Hospitals- Hahnemann, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Lifespan: The Miriam Hospital, Providence, Rhode Island
  - Roger Williams Medical Center/Brown University, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center - Knoxville, Knoxville, Tennessee
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia
  - Virginia Baptist Hospital, Lynchburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Oncology Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
- Canada (16):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - Civic Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Department of Oncology, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Garofalo MC, Winter K, Regine WF, et al.: Recursive partitioning analysis (RPA) of prognostic factors in six Radiation Therapy Oncology Group (RTOG) trials of chemoradiotherapy for unresectable pancreatic cancer. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-144, S80-1, 2006.
- [Result] Konski AA, Winter K, Khor L, et al.: Over-expression of RIa subunit (RIas) of protein kinase A may be a marker for favorable pancreatic cancer: an analysis of patients treated on Radiation Therapy Oncology Group (RTOG) 98-12. [Abstract] American Society of Clinical Oncology 2006 Gastrointestinal Cancers Symposium, 26-28 January 2006, San Francisco, California. A-148, 2006.
- [Result] Rich T, Harris J, Abrams R, Erickson B, Doherty M, Paradelo J, Small W Jr, Safran H, Wanebo HJ. Phase II study of external irradiation and weekly paclitaxel for nonmetastatic, unresectable pancreatic cancer: RTOG-98-12. Am J Clin Oncol. 2004 Feb;27(1):51-6. doi: 10.1097/01.coc.0000046300.88847.bf. PMID 14758134
- [Result] Rich T, Harris J, Abrams R, et al.: A phase II study of external irradiation and weekly paclitaxel for non-metastatic, unresectable pancreatic cancer: a preliminary report of RTOG protocol 98-12. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-51, 29-30, 2001.